CLINICAL TRIAL: NCT06253351
Title: Real-world Use of Hybrid Closed Loop in Adolescents and Young Adults 15-25 Years of Age with Type 1 Diabetes
Acronym: BFHado
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/0060
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Type1 Diabetes; Adolescents; Young Adults
Keywords: type 1 diabetes; hybrid closed-loop; adolescents; young adults; HbA1c; TIR
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group1: Patients between 15 and 25 years old with type 1 diabetes and treated by hybrid closed loop
  Interventions: Device: Hybrid closed loop (HCL)

INTERVENTIONS:
Device: Hybrid closed loop (HCL) — * Control IQ : T-Slim pump with Dexcom G6
  * Smartguard : Medtronic 780G pump with Guardian G4S
  * Diabeloop : Kaliedo pump with Dexcom G6

SUMMARY:
The purpose of this study is to determine the effect of hybrid closed loop on glycemic outcomes in young patients aged between 15 and 25 years old with type 1 diabetes, whatever is their initial metabolic control.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) constitutes a major public health challenge due to acute complications requiring emergency hospitalizations, as well as many chronic complications that need to be managed over the long term. However, these complications can be prevented by maintaining correct glycemic control, according to international guidelines.

For the past few years, the arrival of new technologies as insulin pump and particularly Continuous Glucose Monitoring (CGM) showed a significant improvement on metabolic control.

Nevertheless, adolescents and young adults with type 1 diabetes need a special focus because they still fail to meet glycemic control targets.

At this time, hybrid closed loop, pairing Continuous Glucose Monitoring with insulin pump, enables insulin delivery in a semi-autonomous way thanks to algorithms, and leads to the best metabolic results we've never got in randomized trials and real-world studies.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 15 and 25 years old
* Type 1 diabetes since at least 1 year at the moment of instauring HCL
* At least 3 months of HCL use

Exclusion Criteria:

* Informed patient that have been opposed for their data collect

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Tertiary care center from Centre Hospitalier Sud Francilien
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
HbA1c after HCL | at 3 months
  Comparison of HbA1c (%) before and after HCL (at least 3 months of use)

SECONDARY OUTCOMES:
HbA1c after HCL | at 6 months
  Comparison of HbA1c (%) before and after HCL (at least 3 months of use)
HbA1c after HCL | at 12 months
  Comparison of HbA1c (%) before and after HCL (at least 3 months of use)
HbA1c after HCL | at 24 months
  Comparison of HbA1c (%) before and after HCL (at least 3 months of use)
Use of HCL | at 3 months
  Percentage of use of HCL
HCL stop | at 3 months
  number of HCL stop
Glycemic parameters with CGM | at 3 months
  pourcentage time In Range (TIR) 70-180 mg/dl
Glycemic parameters with CGM | at 3 months
  pourcentage time Below Range (TBR) < 70 mg/dl
Glycemic parameters with CGM | at 3 months
  pourcentage Coefficient of Variation (CV)
keto-acidosis and severe hypoglycemia | at 3 months
  Comparision of keto-acidose and severe hypoglycemia events the year before HCL and after HCL
retinopathy | at 3 months
  Comparison of retinography results before HCL and after HCL
nephropathy | at 3 months
  Comparison microalbuminuria/creatininuria dosage the year before HCL and after HCL

CONTACTS AND LOCATIONS:
Overall Officials: Juliette EROUKHMANOFF, MD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No